CLINICAL TRIAL: NCT04922840
Title: Improved Cardiovascular Health for Patients With Inflammatory Joint Diseases
Acronym: ExeHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Dam Foundation (Other); The Norwegian Rheumatism Association (Other); Norwegian Health Association (Other)
Responsible Party: Principal Investigator, Anne Therese Tveter, Principal Investigator, Assosiate Professor, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/FO347439
Record Dates: First submitted 2021-05-15; First posted 2021-06-11 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Spondyloarthritis; Rheumatoid Arthritis; Psoriatic Arthritis
Keywords: Exercise; Cardiovascular disease; Cardiovascular risk; High-intensity training; Physiotherapy; High-intensity exercise; Inflammatory joint disease
MeSH Terms: conditions — Spondylarthritis; Arthritis, Rheumatoid; Arthritis, Psoriatic; Motor Activity; Cardiovascular Diseases | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will be allocated 1:1 according to a computer-generated randomization scheme, stratified by sex
Who Masked: Investigator
Masking Description: The trial is single-blinded with investigator (KRN) masked for group allocation to reduce risk of bias. Patients are not blinded to treatment exposure nor study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity exercise (HIIT) (Experimental): Usual care; CVD risk assessment, lifestyle advice (heart-healthy diet, regular exercise, weight management and non-smoking) and relevant medication.
  The 12-week intervention is carried out as individual or group sessions with maximal 4 patients, supervised by physiotherapists in primary health care. The HIIT group complete two weekly HIIT sessions and a third weekly session with exercise at moderate intensity. Exercise is tailored to each individual to provide the same relative exercise stress and to ensure progression. Target exercise intensity is tracked by a heart rate monitor.
  Individual exercise session are recorded in a training diary. Succeeding the intervention, a questionnaire will be distributed to patients in the HIIT group. Semi-structured interviews will target physiotherapists supervising HIIT and 5-7 patients in the HIIT group.
  Interventions: Behavioral: High-intensity exercise (HIIT)
- Usual care (No Intervention): Control group participants receive the same treatment as usual care; CVD risk assessment including lifestyle advice (heart-healthy diet, regular exercise, weight management and non-smoking) and relevant medication. Control group participants are invited to a physiotherapist-led theoretical and practical HIIT session following study completion.

INTERVENTIONS:
Behavioral: High-intensity exercise (HIIT) — 12 week intervention: Two weekly sessions of 35-40 min exercise: 10 min warm-up, followed by 4x4 min at 90-95% peak heart rate (HRpeak) interspaced by 2-3 min active breaks at 60-70% HRpeak and a third weekly session with continuous exercise for a minimum of 40 min at moderate intensity.
  Arms: High-intensity exercise (HIIT)

SUMMARY:
Inflammatory joint diseases (IJD) are autoimmune diseases with common symptoms of joint inflammation, pain, stiffness and fatigue. Compared to the general population, this large patient-group has an increased risk of cardiovascular disease (CVD) and CVD-related mortality. Patients with IJD call for improved CVD screening and risk management as well as access to evidence-based non-pharmacological treatment alternatives. Evidence supports high intensity training (HIIT) in mitigating risk of CVD and inflammation, but the evidence of these cardioprotective benefits is unclear in patients with IJD and the feasibility of HIIT protocols in daily clinical care needs to be addressed. Cardiorespiratory fitness (CRF) is an important physiological marker and highly correlated to risk of CVD. Despite strong recommendations, routine assessment of CRF is seldom performed in clinical care.

The ExeHeart study will assess the potential cardioprotective and disease-modifying effect of HIIT in IJD in a randomized controlled trial. Furthermore, the ExeHeart-study will report on the validity of non-exercise measures of cardiorespiratory fitness (eCRF) measures for use in daily clinical care. Additionally, we will explore the feasibility of HIIT by addressing adherence and fidelity to the HIIT treatment protocol in a primary care setting

DETAILED DESCRIPTION:
The study is a two-armed randomized controlled trial (RCT). Patients aged 18-70 years presenting with inflammatory joint disease at the Preventive Cardio-Rheuma clinic at Diakonhjemmet hospital (Oslo) will be included if eligible for the study. Succeeding baseline testing, participants are randomized to either experimental group (high-intensity exercise-HIIT) or control group (usual care).

The research questions are:

1. Is a 12-week HIIT program effective on VO2peak, inflammatory markers and risk of cardiovascular disease in patients with inflammatory joint disease and what is the association between VO2peak and disease-specific and cardiovascular disease-related variables?
2. Is a non-exercise cardio-respiratory fitness algorithm (eCRF) valid in determining longitudinal change in VO2peak in patients with inflammatory joint disease?
3. How feasible is a HIIT intervention in primary care in patients with inflammatory joint disease in terms of adherence and fidelity to the exercise program?

The primary analysis will be a between group comparison of VO2peak levels. This will be carried out according to the intention-to-treat principle, and done by the analysis of covariance (ANCOVA), adjusting for VO2peak values at baseline along with stratification factors used in the randomization. Secondary analyses will include between group comparisons on secondary endpoints, as well as comparisons in the per protocol population. No adjustment for multiple testing will be done.

The association between VO2peak and changes in inflammatory markers, disease activity and CVD risk will be assessed using multiple regression.

The validity of eCRF models to accurately detect longitudinal change in VO2peak from baseline to 3-month and 6-month follow-up will be assessed with Pearson or Spearman correlation by comparing VO2peak derived from a cardiopulmonary exercise test to eCRF.

The feasibility of a HIIT program and adherence will be examined with descriptive statistics. Adherence to the prescribed HIIT intervention will be recorded by attendance to exercise sessions. Quality of treatment delivery will be quantified as the number of exercise sessions complying with the planned exercise intensity and number of exercise sessions requiring dose modifications such as lower exercise intensity or early session termination. At the 3-month timepoint, an electronic questionnaire will be distributed to patients in the HIIT group. Questions regarding feasibility and implementation fidelity will address patients' acceptability and satisfaction with the HIIT program. The ExeHeart study will also include semi-structured interviews, targeting physiotherapists in charge of supervising the exercise sessions and 5-7 patients in the intervention group. The interviews will explore barriers and facilitators in exercise adherence, experience with the protocol and perceived effects of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70
* BMI: 18.5-40
* Inflammatory joint disease verified by physician
* Able to walk unaided and continuously for ≥ 15 min.
* Norwegian or English speaking

Exclusion Criteria:

* Sustained lower extremity injury ≤12 months, including surgery
* Neurological disease
* Absolute contraindication to maximal exercise test
* Cognitive impairment
* Participation in structured high-intensity exercise ≥ 1/week in the last 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen uptake - VO2peak ml/kg/min | 3 months post baseline
  VO2peak, expressed in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min). VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion

SECONDARY OUTCOMES:
Peak oxygen uptake - VO2peak L/min | 3 months post baseline
  VO2peak, expressed in liters per minute. VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion
Peak oxygen uptake - VO2peak ml/kg/min | Baseline
  VO2peak, expressed in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min). VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion (RPE 0-10)
Peak oxygen uptake - VO2peak ml/kg/min | 6 months post baseline
  VO2peak, expressed in milliliters of oxygen per kilogram of body weight per minute (ml/kg/min). VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion (RPE 0-10)
Peak oxygen uptake - VO2peak L/min | Baseline
  VO2peak, expressed in liters per minute. VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion (RPE 0-10)
Peak oxygen uptake - VO2peak L/min | 6 months post baseline
  VO2peak, expressed in liters per minute. VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion (RPE 0-10)
Change in VO2peak (ml/kg/min) from baseline to 3 months past baseline | 3 months post baseline
  Change in VO2peak, expressed in milliliters of oxygen per kilogram of body weight per minute from baseline to 6 months (3 months post intervention) . VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion
Change in VO2peak (ml/kg/min) from baseline to 6 months post baseline | 6 months
  Change in VO2peak, expressed in milliliters of oxygen per kilogram of body weight per minute from baseline to 6 months (3 months post intervention) . VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion
Change in VO2peak L/min from baseline to 3 months post baseline | 3 months post baseline
  VO2peak, expressed in liters per minute(L/min). VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion
Change in VO2peak L/min from baseline to 6 months post baseline | 6 months post baseline
  VO2peak, expressed in liters per minute(L/min). VO2peak will be measured by a Cardiopulmonary Exercise test (CPET) on a treadmill, using electrocardiogram (ECG), breath-by-breath gas analyzing system, blood pressure (BP) monitor, pulse oximetry, and Borg rating of perceived exertion
Body composition | Baseline
  Body scan to estimate total and regional distribution of lean body mass and fat mass
Body composition | 3 months post baseline
  Body scan to estimate total and regional distribution of lean body mass and fat mass
Body composition | 6 months post baseline
  Body scan to estimate total and regional distribution of lean body mass and fat mass
Ventilatory threshold 1 | Baseline
  Point during at which ventilation starts to increase at a faster rate than VO2 - derived from CPET
Ventilatory threshold 1 | 3 months post baseline
  Point during exercise at which ventilation starts to increase at a faster rate than VO2 - derived from CPET
Ventilatory threshold 1 | 6 months post baseline
  Point during exercise at which ventilation starts to increase at a faster rate than volume of oxygen (VO2) - derived from CPET
Ventilatory threshold 2 | Baseline
  The point at which the oxygen demand of the muscles exceeds the ability of the cardiopulmonary system to supply oxygen- derived from CPET
Ventilatory threshold 2 | 3 months post baseline
  The point at which the oxygen demand of the muscles exceeds the ability of the cardiopulmonary system to supply oxygen- derived from CPET
Ventilatory threshold 2 | 6 months post baseline
  The point at which the oxygen demand of the muscles exceeds the ability of the cardiopulmonary system to supply oxygen- derived from CPET
Breathing reserve | Baseline
  Difference between the maximal voluntary ventilation (MVV) and the maximum ventilation measured during CPET
Breathing reserve | 3 months post baseline
  Difference between the maximal voluntary ventilation (MVV) and the maximum ventilation measured during CPET
Breathing reserve | 6 months post baseline
  Difference between the maximal voluntary ventilation (MVV) and the maximum ventilation measured during CPET
Oxygen pulse | Baseline
  The oxygen pulse is the oxygen (O2) divided by heart rate, and represents the product of the stroke volume and the arterial-venous oxygen difference. Derived from CPET.
Oxygen pulse | 3 months post baseline
  The oxygen pulse is the oxygen (O2) divided by heart rate, and represents the product of the stroke volume and the arterial-venous oxygen difference. Derived from CPET.
Oxygen pulse | 6 months post baseline
  The oxygen pulse is the oxygen (O2) divided by heart rate, and represents the product of the stroke volume and the arterial-venous oxygen difference. Derived from CPET.
Ventilatory equivalents for oxygen (VE/VO2) | Baseline
  Ratio of the volume of gas expired per minute to the volume of oxygen consumed per minute- derived from CPET
Ventilatory equivalents for oxygen (VE/VO2) | 3 months post baseline
  Ratio of the volume of gas expired per minute to the volume of oxygen consumed per minute- derived from CPET
Ventilatory equivalents for oxygen (VE/VO2) | 6 months post baseline
  Ratio of the volume of gas expired per minute to the volume of oxygen consumed per minute- derived from CPET
Ventilatory equivalents for carbon dioxide(VE/VCO2) | Baseline
  Ratio of the volume of gas expired per minute to the volume of carbon dioxide produced per minute- derived from CPET
Ventilatory equivalents for carbon dioxide(VE/VCO2) | 3 months post baseline
  Ratio of the volume of gas expired per minute to the volume of carbon dioxide produced per minute- derived from CPET
Ventilatory equivalents for carbon dioxide (VE/VCO2) | 6 months post baseline
  Ratio of the volume of gas expired per minute to the volume of carbon dioxide produced per minute- derived from CPET
Respiratory Exchange Ratio (RER) | Baseline
  Ratio of carbon dioxide output/oxygen uptake (VCO2/VO2) at peak exercise intensity - derived from CPET
Respiratory Exchange Ratio (RER) | 3 months post baseline
  Ratio of carbon dioxide output/oxygen uptake (VCO2/VO2) at peak exercise intensity - derived from CPET
Respiratory Exchange Ratio (RER) | 6 months post baseline
  Ratio of carbon dioxide output/oxygen uptake (VCO2/VO2) at peak exercise intensity - derived from CPET
Blood lactate concentration | Baseline
  Sampled from fingertip within 60 sec of CPET completion to assess level of anaerobic processes
Blood lactate concentration | 3 months post baseline
  Sampled from fingertip within 60 sec of CPET completion to assess level of anaerobic processes
Blood lactate concentration | 6 months post baseline
  Sampled from fingertip within 60 sec of CPET completion to assess level of anaerobic processes
C-Reactive protein | Baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for C-Reactive protein
C-Reactive protein | 3 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for C-Reactive protein
C-Reactive protein | 6 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for C-Reactive protein
Erythrocyte Sedimentation Rate | Baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for Erythrocyte Sedimentation Rate
Erythrocyte Sedimentation Rate | 3 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for Erythrocyte Sedimentation Rate
Erythrocyte Sedimentation Rate | 6 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for Erythrocyte Sedimentation Rate
Total cholesterol | Baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for total cholesterol
Total cholesterol | 3 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for total cholesterol
Total cholesterol | 6 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for total cholesterol
High-density lipoproteins | Baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for high-density lipoproteins
High-density lipoproteins | 3 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for high-density lipoproteins
High-density lipoproteins | 6 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for high-density lipoproteins
Low-density lipoproteins | Baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for low-density lipoproteins
Low-density lipoproteins | 3 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for low-density lipoproteins
Low-density lipoproteins | 6 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for low-density lipoproteins
Triglycerides | Baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for triglycerides
Triglycerides | 3 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for triglycerides
Triglycerides | 6 months post baseline
  Non-fasting blood samples are measured at the hospital laboratory and analysed for triglycerides
Blood pressure | Baseline
  Supine systolic and diastolic blood pressure
Blood pressure | 3 months post baseline
  Supine systolic and diastolic blood pressure
Blood pressure | 6 months post baseline
  Supine systolic and diastolic blood pressure
Body Mass Index | Baseline
  Weight in kilograms divided by the square of height in meters
Body Mass Index | 3 months post baseline
  Weight in kilograms divided by the square of height in meters
Body Mass Index | 6 months post baseline
  Weight in kilograms divided by the square of height in meters
Waist circumference | Baseline
  Waist girth in centimeters. Measured in a standing position after a full exhale.
Waist circumference | 3 months post baseline
  Waist girth in centimeters. Measured in a standing position after a full exhale.
Waist circumference | 6 months post baseline
  Waist girth in centimeters. Measured in a standing position after a full exhale.
Resting heart rate | Baseline
  Recorded in conjunction with blood pressure measurement at rest- resting supine on a bench
Resting heart rate | 3 months post baseline
  Recorded in conjunction with blood pressure measurement at rest- resting supine on a bench
Resting heart rate | 6 months post baseline
  Recorded in conjunction with blood pressure measurement at rest- resting supine on a bench
Health-related quality of life, EuroQoL (EQ5D-5L) | Baseline
  Health-related quality of life is measured by the EQ5D-5L questionnaire. Patients are asked to answer their ability to perform walking, personal care and activities of daily life on a 5 point Likert scale from no difficulties to not able to. Pain and anxiety/depression is measured on a 5 point Likert scale from no pain to very strong pain, and no anxiety/depression to extremely anxious/depressed. General experience of health is measured from 0 (worst health) to 100 (best health) on a numeric rating scale.
Health-related quality of life, EuroQoL (EQ5D-5L) | 3 months post baseline
  Health-related quality of life is measured by the EQ5D-5L questionnaire. Patients are asked to answer their ability to perform walking, personal care and activities of daily life on a 5 point Likert scale from no difficulties to not able to. Pain and anxiety/depression is measured on a 5 point Likert scale from no pain to very strong pain, and no anxiety/depression to extremely anxious/depressed. General experience of health is measured from 0 (worst health) to 100 (best health) on a numeric rating scale.
Health-related quality of life, EuroQoL (EQ5D-5L) | 6 months post baseline
  Health-related quality of life is measured by the EQ5D-5L questionnaire. Patients are asked to answer their ability to perform walking, personal care and activities of daily life on a 5 point Likert scale from no difficulties to not able to. Pain and anxiety/depression is measured on a 5 point Likert scale from no pain to very strong pain, and no anxiety/depression to extremely anxious/depressed. General experience of health is measured from 0 (worst health) to 100 (best health) on a numeric rating scale.
Frequency of medication | Baseline
  Usage of medications last three months. Measured in frequency.
Dosage of medication | Baseline
  Usage of medications last three months. Measured in dosage.
Dosage of medication | 3 months post baseline
  Usage of medications last three months. Measured in dosage
Frequency of medication | 3 months post baseline
  Usage of medications last three months. Measured in frequency
Dosage of medication | 6 months post baseline
  Usage of medications last three months. Measured in dosage.
Frequency of medication | 6 months post baseline
  Usage of medications last three months. Measured in frequency.
Self-reported fatigue | Baseline
  Last week's experience of fatigue is measured on a Numeric rating scale from 0 (No fatigue) to 10 (Worst imaginable fatigue).
Self-reported fatigue | 3 months post baseline
  Last week's experience of fatigue is measured on a Numeric rating scale from 0 (No fatigue) to 10 (Worst imaginable fatigue).
Self-reported fatigue | 6 months post baseline
  Last week's experience of fatigue is measured on a Numeric rating scale from 0 (No fatigue) to 10 (Worst imaginable fatigue).
Self-reported pain | Baseline
  Last week's experience of pain measured by numeric rating scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Self-reported pain | 3 months post baseline
  Last week's experience of pain measured by numeric rating scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Self-reported pain | 6 months post baseline
  Last week's experience of pain measured by numeric rating scale ranging from 0 (no pain) to 10 (worst imaginable pain).
Self-reported physical activity (HUNT) | Baseline
  Measured by questions from the Nord-Trøndelag Health study (HUNT): average frequency (never/<1 per week/1 per week/2-3 per week/almost every day), intensity (easy without losing my breath or breaking into a sweat/so hard that I lose my breath and break into a sweat/I push myself to near-exhaustion) and duration (less than 15 minutes/15-29 minutes/30 minutes to 1 hour/more than 1 hour) of physical activity.
Self-reported physical activity (HUNT) | 3 months post baseline
  Measured by questions from the Nord-Trøndelag Health study (HUNT): average frequency (never/<1 per week/1 per week/2-3 per week/almost every day), intensity (easy without losing my breath or breaking into a sweat/so hard that I lose my breath and break into a sweat/I push myself to near-exhaustion) and duration (less than 15 minutes/15-29 minutes/30 minutes to 1 hour/more than 1 hour) of physical activity.
Self-reported physical activity (HUNT) | 6 months post baseline
  Measured by questions from the Nord-Trøndelag Health study (HUNT): average frequency (never/<1 per week/1 per week/2-3 per week/almost every day), intensity (easy without losing my breath or breaking into a sweat/so hard that I lose my breath and break into a sweat/I push myself to near-exhaustion) and duration (less than 15 minutes/15-29 minutes/30 minutes to 1 hour/more than 1 hour) of physical activity.
SCORE2 | Baseline
  Systemic Coronary Risk Estimation 2 Evaluation: Age, sex, smoking status, non-HDL blood cholesterol and systolic blood pressure is used to estimate 10-year risk of fatal and non-fatal cardiovascular disease.
SCORE2 | 3 months post baseline
  Systemic Coronary Risk Estimation 2 Evaluation: Age, sex, smoking status, non-HDL blood cholesterol and systolic blood pressure is used to estimate 10-year risk of fatal and non-fatal cardiovascular disease.
SCORE2 | 6 months post baseline
  Systemic Coronary Risk Estimation 2 Evaluation: Age, sex, smoking status, non-HDL blood cholesterol and systolic blood pressure is used to estimate 10-year risk of fatal and non-fatal cardiovascular disease.
Forced vital capacity | Baseline
  Volume of air that can be forcefully exhaled after a full inspiration, measured in liters. Obtained from spirometry
Forced vital capacity | 3 months post baseline
  Volume of air that can be forcefully exhaled after a full inspiration, measured in liters- obtained from spirometry
Forced vital capacity | 6 months post baseline
  Volume of air that can be forcefully exhaled after a full inspiration, measured in liters- obtained from spirometry
Forced expiratory volume in 1 second (FEV1) | Baseline
  Volume of air that can be forcefully exhaled in the first second after a full inspiration, measured in liters- obtained by spirometry
Forced expiratory volume in 1 second (FEV1) | 3 months post baseline
  Volume of air that can be forcefully exhaled in the first second after a full inspiration, measured in liters- obtained by spirometry
Forced expiratory volume in 1 second (FEV1) | 6 months post baseline
  Volume of air that can be forcefully exhaled in the first second after a full inspiration, measured in liters- obtained by spirometry
FEV1/FVC ratio | Baseline
  Ratio (%) of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC)
FEV1/FVC ratio | 3 months post baseline
  Ratio (%) of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC)
FEV1/FVC ratio | 6 months post baseline
  Ratio (%) of forced expiratory volume in 1 second (FEV1) to forced vital capacity (FVC)
Forced expiratory flow | Baseline
  Speed of air during the middle part of a forced expiration, intervals at 25%, 50% and 75% of exhaled FVC, measured in liter per second (L/s) - obtained by spirometry
Forced expiratory flow | 3 months post baseline
  Speed of air during the middle part of a forced expiration, intervals at 25%, 50% and 75% of exhaled FVC, measured in liter per second (L/s) - obtained by spirometry
Forced expiratory flow | 6 months post baseline
  Speed of air during the middle part of a forced expiration, intervals at 25%, 50% and 75% of exhaled FVC, measured in liter per second (L/s) - obtained by spirometry
Peak expiratory flow (PEF) | Baseline
  Maximum speed of expiration, expressed in liters per minute (L/min)- obtained from spirometry
Peak expiratory flow (PEF) | 3 months post baseline
  Maximum speed of expiration, expressed in liters per minute (L/min)- obtained from spirometry
Peak expiratory flow (PEF) | 6 months post baseline
  Maximum speed of expiration, expressed in liters per minute (L/min)- obtained from spirometry
Maximum voluntary ventilation (MVV) | Baseline
  Measure of the maximum amount of air that can be inhaled and exhaled in one minute. Measured over a 6- or 12-second time period, extrapolated to a value for one minute, expressed in liters/minute (L/min)- obtained from spirometry
Maximum voluntary ventilation (MVV) | 3 months post baseline
  Measure of the maximum amount of air that can be inhaled and exhaled in one minute. Measured over a 6- or 12-second time period, extrapolated to a value for one minute, expressed in liters/minute (L/min)- obtained from spirometry
Maximum voluntary ventilation (MVV) | 6 months post baseline
  Measure of the maximum amount of air that can be inhaled and exhaled in one minute. Measured over a 6- or 12-second time period, extrapolated to a value for one minute, expressed in liters/minute (L/min)- obtained from spirometry
Psoriatic Arthritis Impact of Disease (PsAID) | Baseline
  Patient-reported outcome measure for assessing psoriatic arthritis. Calculated based on 9 Numerical rating scales (NRS) questions regarding pain, fatigue, skin, work and/or leisure activities, function, discomfort, sleep, coping and anxiety. Each NRS is assessed as a number between 0 and 10. Range of final PsAID value is 0-10 where higher figures indicate worse status. Relevant for study participants with psoriatic arthritis.
Psoriatic Arthritis Impact of Disease (PsAID) | 3 months post baseline
  Patient-reported outcome measure for assessing psoriatic arthritis. Calculated based on 9 Numerical rating scales (NRS) questions regarding pain, fatigue, skin, work and/or leisure activities, function, discomfort, sleep, coping and anxiety. Each NRS is assessed as a number between 0 and 10. Range of final PsAID value is 0-10 where higher figures indicate worse status. Relevant for study participants psoriatic arthritis.
Psoriatic Arthritis Impact of Disease (PsAID) | 6 months post baseline
  Patient-reported outcome measure for assessing psoriatic arthritis. Calculated based on 9 Numerical rating scales (NRS) questions regarding pain, fatigue, skin, work and/or leisure activities, function, discomfort, sleep, coping and anxiety. Each NRS is assessed as a number between 0 and 10. Range of final PsAID value is 0-10 where higher figures indicate worse status. Relevant for study participants with psoriatic arthritis.
Rheumatoid arthritis impact of disease (RAID) | Baseline
  Patient-reported outcome measure for assessing rheumatoid arthritis. Calculated based on 7 Numerical rating scales (NRS) questions regarding pain, functional capacity, fatigue, physical wellbeing, emotional wellbeing, quality of sleep and coping. Each NRS is assessed as a number between 0 and 10. Range of final RAID value is 0-10 where higher figures indicate worse status. Relevant for study participants with rheumatoid arthritis.
Rheumatoid arthritis impact of disease (RAID) | 3 months post baseline
  Patient-reported outcome measure for assessing rheumatoid arthritis. Calculated based on 7 Numerical rating scales (NRS) questions regarding pain, functional capacity, fatigue, physical wellbeing, emotional wellbeing, quality of sleep and coping. Each NRS is assessed as a number between 0 and 10. Range of final RAID value is 0-10 where higher figures indicate worse status. Relevant for study participants with rheumatoid arthritis.
Rheumatoid arthritis impact of disease (RAID) | 6 months post baseline
  Patient-reported outcome measure for assessing rheumatoid arthritis. Calculated based on 7 Numerical rating scales (NRS) questions regarding pain, functional capacity, fatigue, physical wellbeing, emotional wellbeing, quality of sleep and coping. Each NRS is assessed as a number between 0 and 10. Range of final RAID value is 0-10 where higher figures indicate worse status. Relevant for study participants with rheumatoid arthritis.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline
  Patient-reported outcome measure for assessing ankylosing spondylitis. Calculated based on 6 Numerical rating scales (NRS) questions regarding fatigue, pain, spinal pain, joint pain, pain on palpation of areas with localized tenderness, morning stiffness severity and morning stiffness duration. Each NRS is assessed as a number between 0 and 10. Range of final BASDAI value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 3 months post baseline
  Patient-reported outcome measure for assessing ankylosing spondylitis. Calculated based on 6 Numerical rating scales (NRS) questions regarding fatigue, pain, spinal pain, joint pain, pain on palpation of areas with localized tenderness, morning stiffness severity and morning stiffness duration. Each NRS is assessed as a number between 0 and 10. Range of final BASDAI value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 6 months post baseline
  Patient-reported outcome measure for assessing ankylosing spondylitis. Calculated based on 6 Numerical rating scales (NRS) questions regarding fatigue, pain, spinal pain, joint pain, pain on palpation of areas with localized tenderness, morning stiffness severity and morning stiffness duration. Each NRS is assessed as a number between 0 and 10. Range of final BASDAI value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline
  Patient-reported outcome measure for assessing functional limitation in patients with ankylosing spondylitis. Calculated based on 10 Numerical rating scales (NRS) questions, 8 questions regarding functional limitations and 2 questions regarding the ability to cope with everyday life. Each NRS is assessed as a number between 0 and 10. Range of final BASFI value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 3 months post baseline
  Patient-reported outcome measure for assessing functional limitation in patients with ankylosing spondylitis. Calculated based on 10 Numerical rating scales (NRS) questions, 8 questions regarding functional limitations and 2 questions regarding the ability to cope with everyday life. Each NRS is assessed as a number between 0 and 10. Range of final BASFI value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 6 months post baseline
  Patient-reported outcome measure for assessing functional limitation in patients with ankylosing spondylitis. Calculated based on 10 Numerical rating scales (NRS) questions, 8 questions regarding functional limitations and 2 questions regarding the ability to cope with everyday life. Each NRS is assessed as a number between 0 and 10. Range of final BASFI value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Global Score (BAS-G) | Baseline
  Patient-reported outcome measure for assessing ankylosing spondylitis. Calculated based on 2 Numerical rating scales (NRS) questions regarding patients's well-being the previous week and previous six months. Range of final BAS-G value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Global Score (BAS-G) | 3 months post baseline
  Patient-reported outcome measure for assessing ankylosing spondylitis. Calculated based on 2 Numerical rating scales (NRS) questions regarding patients's well-being the previous week and previous six months. Range of final BAS-G value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Bath Ankylosing Spondylitis Global Score (BAS-G) | 6 months post baseline
  Patient-reported outcome measure for assessing ankylosing spondylitis. Calculated based on 2 Numerical rating scales (NRS) questions regarding patients's well-being the previous week and previous six months. Range of final BAS-G value is 0-10 where higher figures indicate worse status. Relevant for study participants with spondyloarthritis.
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 3 months post baseline
  Composite score to assess disease activity in ankylosing spondylitis. Calculated based on three questions from BASDAI, patient global assessment on 0-10 scale and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with spondyloarthritis.
Ankylosing Spondylitis Disease Activity Score (ASDAS) | 6 months post baseline
  Composite score to assess disease activity in ankylosing spondylitis. Calculated based on three questions from BASDAI, patient global assessment on 0-10 scale and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with spondyloarthritis.
Ankylosing Spondylitis Disease Activity Score (ASDAS) | Baseline
  Composite score to assess disease activity in ankylosing spondylitis. Calculated based on three questions from BASDAI, patient global assessment on 0-10 scale and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with spondyloarthritis.
Disease Activity Score Calculator for Rheumatoid Arthritis (DAS28) | Baseline
  Composite score to assess disease activity in rheumatoid arthritis. Calculated based on number of swollen (0-28) and tender joints (0-28), patient global assessment of health and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with rheumatoid arthritis.
Disease Activity Score Calculator for Rheumatoid Arthritis (DAS28) | 3 months post baseline
  Composite score to assess disease activity in rheumatoid arthritis. Calculated based on number of swollen (0-28) and tender joints (0-28), patient global assessment of health and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with rheumatoid arthritis.
Disease Activity Score Calculator for Rheumatoid Arthritis (DAS28) | 6 months post baseline
  Composite score to assess disease activity in rheumatoid arthritis. Calculated based on number of swollen (0-28) and tender joints (0-28), patient global assessment of health and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with rheumatoid arthritis.
Disease Activity in PSoriatic Arthritis (DAPSA) | Baseline
  Composite score to assess disease activity in psoriatic arthritis. Calculated based on number of swollen (0-66) and tender joints (0-68), patient global assessment of health and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with psoriatic arthritis
Disease Activity in PSoriatic Arthritis (DAPSA) | 3 months post baseline
  Composite score to assess disease activity in psoriatic arthritis. Calculated based on number of swollen (0-66) and tender joints (0-68), patient global assessment of health and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with psoriatic arthritis
Disease Activity in PSoriatic Arthritis (DAPSA) | 6 months post baseline
  Composite score to assess disease activity in psoriatic arthritis. Calculated based on number of swollen (0-66) and tender joints (0-68), patient global assessment of health and C-Reactive Protein or Erythrocyte Sedimentation Rate from blood samples. Relevant for study participants with psoriatic arthritis
Post-exercise questionnaire | 3 months post baseline
  Electronic questionnaire distributed to patients in the experimental group upon completion of HIT intervention. 14 statements related to participation in the HIT exercise intervention and perceived intensity, duration and frequency of the exercise intervention. Scored on a 5 point Likert scale ranging from strongly disagree to strongly agree.
Use of healthcare services | Baseline
  Use of health care services is measured by number of consultations to general practitioner, medical specialist, physiotherapist, occupational therapist, Healthy Life Centres, psychologist in the last three months.
Use of healthcare services | 3 months post baseline
  Use of health care services is measured by number of consultations to general practitioner, medical specialist, physiotherapist, occupational therapist, Healthy Life Centres, psychologist in the last three months.
Use of healthcare services | 6 months post baseline
  Use of health care services is measured by number of consultations to general practitioner, medical specialist, physiotherapist, occupational therapist, Healthy Life Centres, psychologist in the last three months.
Smoking status | Baseline
  Registered by self-report; I smoke daily, I am a former smoker , I have never smoked
Smoking status | 3 months post baseline
  Registered by self-report; I smoke daily, I am a former smoker , I have never smoked
Smoking status | 6 months post baseline
  Registered by self-report; I smoke daily, I am a former smoker , I have never smoked
Snuff status | Baseline
  Registered by self-report; I use snuff daily, I have previously used snuff, I have never used snuff
Snuff status | 3 months post baseline
  Registered by self-report; I use snuff daily, I have previously used snuff, I have never used snuff
Snuff status | 6 months post baseline
  Registered by self-report; I use snuff daily, I have previously used snuff, I have never used snuff
Peak heart rate | Baseline
  Peak heart rate observed during CPET
Peak heart rate | 3 months post baseline
  Peak heart rate observed during CPET
Peak heart rate | 6 months post baseline
  Peak heart rate observed during CPET
Augmentation index | Baseline
  Indicator of arterial stiffness, measured by mobil-o-graph at the same time as measure of blood pressure
Augmentation index | 3 months post baseline
  Indicator of arterial stiffness, measured by mobil-o-graph at the same time as measure of blood pressure
Augmentation index | 6 months post baseline
  Indicator of arterial stiffness, measured by mobil-o-graph at the same time as measure of blood pressure
Pulse Wave Velocity | Baseline
  Measure of arterial stiffness- rate at which blood propagates through the vessels. Measured by moil-o-graph at the same time as measure of blood pressure
Pulse Wave Velocity | 3 months post baseline
  Measure of arterial stiffness- rate at which blood propagates through the vessels. Measured by moil-o-graph at the same time as measure of blood pressure
Pulse Wave Velocity | 6 months post baseline
  Measure of arterial stiffness- rate at which blood propagates through the vessels. Measured by moil-o-graph at the same time as measure of blood pressure
Exercise self-efficacy | Baseline
  Measured by Exercise Beliefs and Exercise Habits questionnaire: comprises 20 items addressing exercise self-efficacy (4 items), barriers to exercise (3 items), benefits of exercise (5 items), and impact of exercise on arthritis (8 items), scored on a 5-point Likert scale ranging from strongly disagree to strongly agree. The scores on each subscale is summed up where higher scores indicate better self-efficacy.
Exercise self-efficacy | 3 months post baseline
  Measured by Exercise Beliefs and Exercise Habits questionnaire: comprises 20 items addressing exercise self-efficacy (4 items), barriers to exercise (3 items), benefits of exercise (5 items), and impact of exercise on arthritis (8 items), scored on a 5-point Likert scale ranging from strongly disagree to strongly agree. The scores on each subscale is summed up where higher scores indicate better self-efficacy.
Exercise self-efficacy | 6 months post baseline
  Measured by Exercise Beliefs and Exercise Habits questionnaire: comprises 20 items addressing exercise self-efficacy (4 items), barriers to exercise (3 items), benefits of exercise (5 items), and impact of exercise on arthritis (8 items), scored on a 5-point Likert scale ranging from strongly disagree to strongly agree. The scores on each subscale is summed up where higher scores indicate better self-efficacy.
Exercise frequency | 3 months post baseline
  Participants in the experimental group are asked to record individual exercise session in a training diary. Exercise frequency is recorded.
Exercise intensity | 3 months post baseline
  Participants in the experimental group are asked to record individual exercise session in a training diary. Exercise intensity is recorded by use of a herat rate monitor.
Exercise duration | 3 months post baseline
  Participants in the experimental group are asked to record individual exercise session in a training diary. Exercise duration is recorded.
Early session termination | 3 months post baseline
  Participants in the experimental group are asked to record individual exercise session in a training diary. Early session termination is recorded.
Exercise-related adverse events | 3 months post baseline
  Participants in the experimental group are asked to record individual exercise session in a training diary. Exercise-related adverse events are recorded.
Self-reported cardiovascular health and symptoms | Baseline
  13 yes/no questions regarding self-report of cardiovascular disease, symptoms and cardiac surgery. If the participant answers yes to preliminary question regarding angina, 5 ancillary questions pertaining to angina symptomatology are provided
Self-reported cardiovascular health and symptoms | 3 months post baseline
  13 yes/no questions regarding self-report of cardiovascular disease, symptoms and cardiac surgery. If the participant answers yes to preliminary question regarding angina, 5 ancillary questions pertaining to angina symptomatology are provided
Self-reported cardiovascular health and symptoms | 6 months post baseline
  13 yes/no questions regarding self-report of cardiovascular disease, symptoms and cardiac surgery. If the participant answers yes to preliminary question regarding angina, 5 ancillary questions pertaining to angina symptomatology are provided
Self-report change in physical fitness | 3 months post baseline
  Patient global change in self-perceived physical fitness measured on a 5-point Likert scale ranging from much better to much worse
Self-report change in physical fitness | 6 months post baseline
  Patient global change in self-perceived physical fitness measured on a 5-point Likert scale ranging from much better to much worse
Self-report exercise habits | 3 months post baseline
  Questionnaire; self-report of exercise habits from baseline to 3 months post baseline: Participation in regular exercise (yes/no), if yes: frequency (1-2 times/week, 3-4 times/week, 5 times or more/week) and mode of exercise (endurance exercise, strength exercise, mobility exercise and/or other).
  These questions are only forwarded to participants in the control group at this timepoint. Exercise habits form baseline to 3 months post baseline is recorded via the training diary for participants allocated to HIIT (experimental group): see outcome 153-157.
Self-report exercise habits | 6 months post baseline
  Questionnaire; self-report of exercise habits from 3 months post baseline to 6 months post-baseline: Participation in regular exercise (yes/no), if yes: frequency (1-2 times/week, 3-4 times/week, 5 times or more/week) and mode of exercise (endurance exercise, strength exercise, mobility exercise and/or other).
  These questions are forwarded to all study participants at this timepoint.
Corona virus 19 infection | 3 months post baseline
  Questionnaire; self-report regarding corona virus 19 infection (yes/no, if yes: hospitalization/no hospitalization) from baseline to 3 months post baseline
Corona virus 19 infection | 6 months post baseline
  Questionnaire; self-report regarding corona virus 19 infection (yes/no, if yes: hospitalization/no hospitalization) from 3 months post baseline to 6 montsh post baseline
Corona virus 19 quarantine | 3 months post baseline
  Questionnaire; self-report regarding corona virus 19 quarantine (yes/no) from baseline to 3 months post baseline
Corona virus 19 quarantine | 6 months post baseline
  Questionnaire; self-report regarding corona virus 19 quarantine (yes/no) from 3 months post baseline to 6 months post baseline
Maximum minute ventilation at peak exercise (VEmax, L/min) | Baseline
  Maximum ventilation, recorded from CPET at peak exercise
Maximum minute ventilation at peak exercise (VEmax, L/min) | 3 months post baseline
  Maximum ventilation, recorded from CPET at peak exercise
Maximum minute ventilation at peak exercise (VEmax, L/min) | 6 months post baseline
  Maximum ventilation, recorded from CPET at peak exercise

CONTACTS AND LOCATIONS:
Overall Officials: Anne Therese Tveter, PhD, Principal Investigator — National Resource Center for Rehabilitation in Rheumatology
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Data may be made available upon sound request to the principal investigator

REFERENCES:
- [Derived] Norden KR, Semb AG, Dagfinrud H, Hisdal J, Sexton J, Fongen C, Bakke E, Odegard S, Skandsen J, Blanck T, Metsios GS, Tveter AT. Effect of high-intensity interval training in physiotherapy primary care for patients with inflammatory arthritis: the ExeHeart randomised controlled trial. RMD Open. 2024 Jan 18;10(1):e003440. doi: 10.1136/rmdopen-2023-003440. PMID 38242550
- [Derived] Norden KR, Semb AG, Dagfinrud H, Hisdal J, Odegard S, Sexton J, Fongen C, Skandsen J, Blanck T, Metsios GS, Tveter AT. Associations between cardiovascular risk factors, disease activity and cardiorespiratory fitness in patients with inflammatory joint disease: a cross-sectional analysis. BMC Sports Sci Med Rehabil. 2023 Apr 21;15(1):63. doi: 10.1186/s13102-023-00678-4. PMID 37085935
- [Derived] Norden KR, Dagfinrud H, Semb AG, Hisdal J, Viktil KK, Sexton J, Fongen C, Skandsen J, Blanck T, Metsios GS, Tveter AT. Effect of high-intensity exercise on cardiorespiratory fitness, cardiovascular disease risk and disease activity in patients with inflammatory joint disease: protocol for the ExeHeart randomised controlled trial. BMJ Open. 2022 Feb 17;12(2):e058634. doi: 10.1136/bmjopen-2021-058634. PMID 35177467
- See also: Effect of high-intensity exercise on cardiorespiratory fitness, cardiovascular disease risk and disease activity in patients with inflammatory joint disease: protocol for the ExeHeart randomised controlled trial — https://bmjopen.bmj.com/content/bmjopen/12/2/e058634.full.pdf

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT04922840/SAP_001.pdf